CLINICAL TRIAL: NCT05111587
Title: Epidemiology of Injuries Caused by the Practice of Artificial Structure Climbing: Prospective Cohort Study in Réunion Island
Brief Title: Epidemiology of Injuries Caused by the Practice of Artificial Structure Climbing
Acronym: EPITRAUMABLOC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/27
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Sport Injury
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Participant must complete a questionnaire about injury during climbing practice in an artificial structure

SUMMARY:
This study aims to precisely describe epidemiology of injuries than occur during practice of climbing in artificial structure.

Each participant will complete questionnaires in order to identify injuries. The first questionnaire will be completed at the moment of the inclusion and the second questionnaire will be completed if participant has injuries every 3 months until month 12.

ELIGIBILITY:
Inclusion Criteria:

- person who practices artificial structure climbing

Exclusion Criteria:

* person who refuses to participate
* person under tutorship or curatorship
* person who cannot read and write
* person who wants to leave Reunion Island within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult who practices climbing in artificial structure must be included in Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
location of injury | at month 3
laterality of injury | at month 3
mechanism of injury | at month 3
  it will be identified as a traumatic injury or an overuse. Traumatic injury is due to an acute identified event. An overuse is due to repetitive train injury.
circumstance of injury occurence | at month 3
injury relapse or not | at month 3
  injury relapse is classified as early relapse if occurs within 2 months after the healing, as late relapse if occurs from 2 months to 12 months after the healing or as very late relapse if occurs after more 12 months.
diagnosis of injury | at month 3
  diagnosis will be claissified according to the OSICS 10 classification
record of exposure to injury | at month 3
  Training volume will be recorded by level of practice (leisure practice, club practice and competition practice)

CONTACTS AND LOCATIONS:
Locations (1):
- Climbing structure, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No